CLINICAL TRIAL: NCT03237832
Title: A Phase 1, Single-Center, Randomized, Double-Blind, Placebo-Controlled Safety, Tolerability, and Pharmacokinetic Study of Single Ascending Oral Doses of ARN-6039 in Healthy Adult Subjects.
Brief Title: A Phase 1 Study of ARN-6039
Acronym: ARN-6039
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrien Pharmaceuticals (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: ARN-CLN-0001
Record Dates: First submitted 2017-07-21; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Determine safety and tolerability of ARN-6039 ascending doses compared to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacist preparing the doses was unblended and was responsible for all drug accountability issues, including preparing, labeling, and dispensing study drug according to the randomization code provided. The unblinded pharmacists were responsible for maintaining the blind, consistent with protocol design, throughout the study. All documentation was filed in the Pharmacy Manual, and access to this manual was restricted to the unblinded pharmacists. The subjects, Principal Investigator, and all other personnel involved with subject assessments were blinded to the actual treatment assignments of the subjects (ARN-6039 or placebo) during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Placebo Comparator): Cohort 1 (sentinel group): 1 subject received 50 mg ARN-6039 and 1 subject placebo Cohort 1: 7 subjects received 50 mg ARN-6039 and 1 subject placebo
  Interventions: Drug: ARN-6039; Other: Placebo
- Cohort 2 (Placebo Comparator): Cohort 2 (sentinel group): 1 subject received 100 mg ARN-6039 and 1 subject placebo Cohort 2: 7 subjects received 100 mg ARN-6039 and 1 subject placebo
  Interventions: Drug: ARN-6039; Other: Placebo
- Cohort 3 (Placebo Comparator): Cohort 3 (sentinel group): 1 subject received 150 mg ARN-6039 and 1 subject placebo Cohort 3: 7 subjects received 150 mg ARN-6039 and 1 subject placebo
  Interventions: Drug: ARN-6039; Other: Placebo
- Cohort 4 (Placebo Comparator): Cohort 4 (sentinel group): 1 subject received 200 mg ARN-6039 and 1 subject placebo Cohort : 7 subjects received 200 mg ARN-6039 and 1 subject placebo
  Interventions: Drug: ARN-6039; Other: Placebo
- Cohort 5 (Placebo Comparator): Cohort 5 Period 1, fasted (sentinel group): 1 subject received 300 mg ARN-6039 and 1 subject placebo Cohort 5 Period 1, fasted: 7 subjects received 300 mg ARN-6039 and 1 subject placebo Cohort 5 Period 2, fed (sentinel group): 1 subject received 300 mg ARN-6039 and 1 subject placebo Cohort 5 Period 2, fed: 7 subjects received 300 mg ARN-6039 and 1 subject placebo
  Interventions: Drug: ARN-6039; Other: Placebo

INTERVENTIONS:
Drug: ARN-6039 — Ascending doses per Cohort
Other: Placebo — Placebo to match ARN-6039

SUMMARY:
This Phase 1 study intends to determine the safety and tolerability of ARN-6039 in healthy subjects.

DETAILED DESCRIPTION:
To determine the safety and tolerability in healthy subjects, ARN-6039 will be dosed in a single-center, randomized, double-blind, placebo-controlled, ascending dose study. Five cohorts of 10 subjects will be dosed in ascending order, beginning with a single dose of 50 mg of ARN-6039. Subsequent cohorts will be administered single doses of 100 mg, 150 mg, 200 mg, or 300 mg. Safety, tolerability, and pharmacokinetics will be evaluated prior to each dose escalation using the assessment of all available safety and pharmacokinetic data.

In Cohorts 1 through 4, subjects will receive a single dose of ARN-6039 or matching placebo under fasted conditions. In Cohort 5, subjects will be administered a single dose of ARN-6039 or a single dose of matching placebo under fasted conditions in Period 1 and under fed conditions in Period 2 with a minimum 5-day washout period between each dose.

To support the administration of ARN-6039 in humans, preclinical toxicology studies performed in rats and dogs demonstrated tolerability exceeding the intended therapeutic dose. In addition, the safety and efficacy of ARN-6039 has been demonstrated in model systems and is anticipated to be well tolerated in humans. This study will be the first administration of ARN-6039 in human subjects.

ELIGIBILITY:
Inclusion Criteria:

Only volunteers who met all of the following criteria were included as study subjects:

* Male or female between 18 and 50 years of age, inclusive.
* Female subjects were not pregnant or lactating.
* Female subjects were postmenopausal (at least 2 years prior to dosing) or surgically sterile. Subjects who claimed postmenopausal status had their status confirmed with a follicle-stimulating hormone (FSH) test. Surgically sterile was defined as: Bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months prior to dosing; or Permanent sterilization (e.g., ESSURE procedure) at least 3 months prior to dosing.
* Subjects had a body mass index (BMI) between 19 and 30 kg/m2 (inclusive) and weighed a minimum of 50 kg (110 lbs).
* Subjects voluntarily consented to participate in this study and provided their written informed consent prior to start of any study-specific procedures.
* Subject was willing and able to comply with all trial requirements.
* Subject was willing and able to remain in the study unit for the entire duration of the confinement period and return for an outpatient visit 7 days after study treatment administration.
* Subject's vital signs (measured sitting after 5 minutes rest) at screening were within the following ranges: heart rate: 40-100 beats per minute [bpm]; systolic blood pressure (BP): 90-145 mmHg; diastolic BP: 50-95 mmHg. Out-of-range vital signs could be repeated once. Predose vital signs were assessed by the Principal Investigator or designee (e.g., a medically qualified Sub-Investigator) prior to study drug administration. The Principal Investigator or designee verified the eligibility of each subject with out-of-range vital signs and documented approval prior to dosing.
* Subjects had results within normal range on the following hematology tests performed at screening: hemoglobin, hematocrit, total and differential leukocyte count, and platelet count.
* Subject had results that did not exceed the upper limit of normal range on the following liver function tests performed at screening: aspartate transaminase (AST), alanine transaminase (ALT), and total bilirubin.
* If enrolled in Cohort 5 (the food-effect cohort), subject was willing and able to consume the entire high-calorie, high-fat breakfast meal in the designated timeframe required during the fed period.

Exclusion Criteria:

Volunteers who presented any of the following criteria were excluded as study subjects:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal (including cholecystectomy), endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would likely have interfered with the absorption, disposition, metabolism, or excretion of the investigational product, or would have jeopardized the safety of the subject or the validity of the study results.
* History of cancer with the exception of basal cell carcinoma or squamous cell (skin) carcinoma.
* History of seizure (including febrile seizure) or loss of consciousness.
* History of drug or alcohol abuse or dependence (based on the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition criteria) within the past 2 years.
* Donated blood or plasma or experienced significant loss of blood within 8 weeks prior to admission to the clinic, or planned to donate blood within 1 month after study participation.
* Had a clinically significant abnormal finding on the physical exam, medical history, ECG, or clinical laboratory results at screening.
* Had smoked or used tobacco or nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, etc.) within 30 days prior to the first dose of study medication.
* History or presence of allergic or adverse response to ARN-6039 or related drugs or its excipients.
* Had been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
* Had participated in another clinical trial (randomized subjects only) within 30 days (or 5 half-lives of the investigational product) prior to the first dose of study medication.
* Had used any over-the-counter (OTC) medication, nutritional or dietary supplements, or herbal preparations, (other than acetaminophen and/or multivitamins [acetaminophen 2 grams/day and multivitamins were allowed up to 48 hours prior to dosing]), within 7 days prior to the first dose of medication.
* Had used any prescription medication, except hormonal replacement therapy, within 14 days prior to the first dose of study medication.
* Consumed the following beverages or products within the specified time frame prior to admission to the clinic: Alcohol, grapefruit, Seville oranges (marmalade), xanthine, or quinine within 72 hours; or Caffeine or poppy seeds within 48 hours.
* Had been treated with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) enzymes such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication and that in the Investigator's judgment may have impacted subject safety or the validity of the study results.
* Had a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates) or cotinine.
* Had a positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at screening or had been previously treated for hepatitis B, hepatitis C, or HIV infection.
* Was, for any reason, deemed by the investigator to be inappropriate for this study, including subjects who were unable to communicate or cooperate with the investigator or designee.
* Female with a positive pregnancy test result.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2016-10-06 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in clinical tests results over time | Days -1, 1, 2, 3, and 7
  Assess the results of analytical hematology, serology, and urine tests compared to normal results from baseline to 7 days post administration
Change in vital signs over time | Days -1, 1, 2, 3, and 7
  Assess subject vital signs compared to normal results from baseline to 7 days post administration
Change in physical assessment over time | Days -1, 1, 2, 3, and 7
  Assess results of subject physical examination compared to normal results from baseline to 7 days post administration
Change in electrocardiograms (ECGs) over time | Days -1, 1, 2, 3, and 7
  Assess results of subject electrocardiograms compared to normal from baseline to 7 days post administration
Determine the incidence of Treatment Adverse Events (AEs) over time | Days -1, 1, 2, 3, and 7
  Assess any adverse events compared to normal from baseline to 7 days post administration

SECONDARY OUTCOMES:
Assay maximum plasma concentration (Cmax) over time | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36 and 48 hours after dosing
  Assess the results of the maximum plasma concentration (Cmax) over time in both the unfed and fed state
Assay the time to Cmax (tmax) over time | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36 and 48 hours after dosing
  Assess the results of the assay time to Cmax (tmax) over time in both the unfed and fed state
Assay the area under the plasma concentration time curve from zero to the last measurable concentration (AUC0-t) over time | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36 and 48 hours after dosing
  Assess the results of the assay of the area under the plasma concentration time curve from zero to the last measurable concentration (AUC0-t) over time in both the unfed and fed state
Assay the terminal half-life (t1/2) over time | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36 and 48 hours after dosing
  Assess the results of the assay the terminal half-life (t1/2) over time in both the unfed and fed state
Assay the area under the plasma concentration time curve from zero to infinity (AUC0-inf) over time | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36 and 48 hours after dosing
  Assess the results of the area under the plasma concentration time curve from zero to infinity (AUC0-inf) over time in both the unfed and fed state
Assay the apparent oral clearance (CL/F) over time | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36 and 48 hours after dosing
  Assess the results of the apparent oral clearance (CL/F) over time in both the unfed and fed state

OTHER OUTCOMES:
Identify possible metabolites of ARN-6039. | 7 days +/- 1 day
  Urine was measured using LC-MS/MS to identify ARN-6039 and/or metabolites.

IPD SHARING:
Plan to Share IPD: Yes
This is a single-center, randomized, ascending dose study in which 5 cohorts of healthy male and female subjects will be administered single doses of ARN 6039 or matching placebo; subjects will be blinded to treatment (ARN-6039 vs. placebo). The ARN 6039 dose will be escalated in each cohort. Each individual participant data is available from sponsor company for review.
Supporting Information: CSR
Time Frame: Clinical study report currently available.
Access Criteria: Please contact Dr. Hari Vankayalapati at Arrien Pharmaceuticals LLC (e-mail: hari@arrienpharma.com).